CLINICAL TRIAL: NCT04117074
Title: A Non-Inferiority Randomized Trial Comparing the Impact of Thoracic Epidural Analgesia Versus Surgical Site Infiltration With Liposomal Bupivicaine on the Postoperative Recovery of Patients Following Open Gynecologic Surgery
Brief Title: Thoracic Epidural Analgesia vs Surgical Site Infiltration With Liposomal Bupivacaine Following Open Gynecologic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J17157; IRB00223229 (Other: JHM IRB)
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Surgery; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Tea; Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Thoracic Epidural Analgesia with bupivicaine (Experimental): Thoracic epidural analgesia (TEA): 0.125 % Bupivicaine infusion (5-7 milliliter [mL] per hour) intraoperatively with a 3 mL bolus at the end of the operative procedure just prior to emergence from general anesthesia. Postoperatively 0.0625% Bupivicaine until patient-controlled epidural analgesia (PCEA) pump. PCEA pump 0.0625% bupivacaine at 5-7 mL per hour infusion with a 3 mL q20 minutes demand. PCEA discontinuation with oral tolerance.
  Interventions: Other: Thoracic epidural analgesia (bupivacaine)
- Arm 2: Surgical Site Infiltration with Liposomal Bupivacaine (Experimental): Liposomal bupivacaine (LB) surgical site infiltration: A single 20 mL liposomal bupivacaine vial containing 266 mg of free-base bupivacaine will be mixed with 60 mL of 0.25% bupivacaine hydrochloride (HCl) and then diluted in preservative-free sterile 0.9% saline for maximal volume not to exceed 300 mL. Dilution with 0.9% saline will be dependent upon length of surgical incision per protocol. The solution will be injected using 22-gauge needle in equal distribution into the peritoneum, along the fascia and into the subcutaneous tissues of the surgical wound by trained faculty surgeons.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Surgical site infiltration with 20 mL liposomal bupivacaine prior to laparotomy closure.
  Other Names: Exparel
  Arms: Arm 2: Surgical Site Infiltration with Liposomal Bupivacaine
Other: Thoracic epidural analgesia (bupivacaine) — Perioperative bupivacaine based thoracic epidural placed preoperatively.
  Arms: Arm 1: Thoracic Epidural Analgesia with bupivicaine

SUMMARY:
The goal of this study is to test the hypothesis that surgical site infiltration with liposomal bupivacaine (LB) is non-inferior to and more cost effective than thoracic epidural analgesia (TEA) for patients undergoing open gynecologic surgery on an established enhanced recovery program (ERP) using a non-inferiority randomized trial design. The impact of TEA and surgical site infiltration with LB on neuroendocrine and inflammatory mediators of surgical stress response (SSR) will also be investigated as a translational endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years of age
* Planned laparotomy by the gynecologic oncology service at the sponsor institution.

Exclusion Criteria:

* Individuals who have a contraindication to thoracic epidural analgesia
* Individuals with a coagulation disorder
* Individuals with an infection at the site of epidural placement
* Individuals with intracranial pathology such as non-communicating increased intracranial pressure or obstruction of cerebrospinal fluid flow related to mass lesions
* Individuals with spinal pathology: abnormal spine anatomy, surgical fusion, or spinal column lesions
* Individuals who have a contraindication to liposomal bupivacaine
* Individuals with a known allergic reaction to liposomal bupivacaine
* Individuals with Childs-Pugh Class B or C liver disease
* Individuals who have a history of long-term opioid use for chronic pain, defined as use of opioid pain medications for ≥4 weeks prior to surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Analgesia as assessed by pain intensity scores on a visual analog scale | 0 to 48 hours postoperatively
  Pain intensity will be measured using visual analog scale (VAS) pain intensity scores. The VAS scores pain intensity on a scale of 0-10, where 0 is no pain and 10 is the most severe pain.
Total opioid consumption | 0 to 48 hours postoperatively
  Total opioid consumption in IV mg morphine equivalents from 0 to 48 hours postoperatively will be compared between the two arms.

SECONDARY OUTCOMES:
Change in Patient-perceived quality of recovery as assessed by the Quality of Recovery-15 instrument (QoR-15) | Days 1 through 7 post-intervention
  Mean patient-perceived quality of recovery scores using the Quality of Recovery-15 instrument (QoR-15) on postoperative days 1 to 7 will be compared between the two arms. The QoR-15 is a validated instrument designed to measure the major domains of postoperative recovery including functional independence, physical comfort/pain, psychological/emotional well-being, cognition and satisfaction with a score of 0 indicating the poorest patient-perceived quality of recovery and 150 indicating the highest patient-perceived quality of recovery.
Time (days) to return of bowel function (ROBF) | Up to 7 days post-intervention
  Time to ROBF is defined as the time lapse from the day of surgery (DOS) to the day oral intake is consistently tolerated for 48 hours without vomiting.
Number of participants with postoperative ileus | Up to 7 days post-intervention
  Ileus is defined as the occurrence of postoperative nausea and vomiting requiring cessation of oral intake and initiation of intravenous hydration +/- nasogastric tube placement following documented ROBF or the persistence of these symptoms beyond postoperative day 5 in the absence of ROBF.
Mobility as assessed by the Johns Hopkins Highest Level of Mobility (JH-HLM) scale | Up to 7 days post-intervention
  The Johns Hopkins Highest Level of Mobility scale is an ordinal scale from 1 to 8, with numbers representing mobility milestones that patients accomplish, based on observation. Patients who score a 2 have some type of bed mobility, while those scoring an 8 can walk more than 250 feet.
Degree of sedation as assessed by the Pasero Opioid-Induced Sedation Scale | Up to 7 days post-intervention
  The Pasero Opioid-induced Sedation Scale (POSS) is a valid, reliable tool used to assess sedation when administering opioid medications to manage pain. It uses an ordinal scale of 1-4 with a POSS of 1 or 2 indicating an acceptable level of sedation and a score of 3 or 4 indicating over-sedation and the need for intervention, such as the administration of a reversal agent in the case of a score of 4.
Length of stay | Up to 1 year
  The duration of the index inpatient postoperative admission in days.
Time to postoperative diuresis | Arrival in recovery through hospital discharge, up to 1 year
  Time to diuresis is defined as the recovery time in hours to achieve a net negative fluid balance sustained over a 24 hour time period.
Total intravenous fluids administered in mL | Arrival in recovery through hospital discharge, up to 1 year
Amount of Vasopressor required | Start of operation through hospital discharge, up to 1 year
  Total amount (micrograms) of vasopressor required.
Duration of Vasopressor administration | Start of operation through hospital discharge, up to 1 year
  Duration (minutes) of vasopressor administration.
Number of postoperative complications | Day of admission through postoperative day 30
  Number of postoperative complications (Maryland Hospital Acquired Conditions).
Total direct cost of TEA placement and LB surgical site infiltration | Up to 1 year
  Pharmacy and equipment costs, professional fees and the dollar-value of total OR time required for administration of each intervention will be compared.
Post-discharge narcotic utilization | Postoperative day 14
  Patient reported total outpatient narcotic use in IV morphine (mg) equivalents on nurse phone survey administered on postoperative day 14.
Change in Serum adrenocorticotropic hormone (ACTH) | Baseline and postoperative day 7
  Serum ACTH level in pg/mL.
Change in Epinephrine level (pg/mL) | Baseline and postoperative day 7
Change in Total cortisol level (microgram/dL) | Baseline and postoperative day 7
Change in Anti-diuretic hormone (ADH) level | Baseline and postoperative day 7
  ADH level in pg/mL.
Change in Interleukin-6 level (pg/mL) | Baseline and postoperative day 7
Change in Atrial natriuretic peptide (ANP) level | Baseline and postoperative day 7
  ANP level in pg/mL.
Change in Syndecan-1 level (pg/mL) | Baseline and postoperative day 7
Change in Glycosaminoglycans level (ng/mL) | Baseline and postoperative day 7
Change in Endothelial glycocalyx constituents (ng/mL) | Baseline and postoperative day 7
Change in C-reactive protein level (ng/mL) | Baseline and postoperative day 7
Change in Tumor necrosis factor alpha (TNF-α) level | Baseline and postoperative day 7
  TNF-α level in pg/mL.
Change in Salivary cortisol (microgram/dL) level | Baseline and postoperative day 7
Rate of 30-day hospital readmission | Up to 30 days post discharge from index admission
  Rate of 30-day hospital readmission assessed as the number of participants who get readmitted within 30 days of discharge from the initial admission.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Stone, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No